CLINICAL TRIAL: NCT00320463
Title: Compare Immunogenicity & Reactogenicity of 2 Formulations of GSK Biologicals' DTPa-HBV-IPV/Hib Vaccine (New vs Current) Given in Healthy Infants. The DTPa-HBV-IPV Vaccine (New Formulation) Will Also be Assessed in a 3rd Group of Subjects
Brief Title: Compare Immunogenicity & Safety of 2 Formulations of GSK Biologicals' DTPa-HBV-IPV/Hib Vaccine Given in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 105910
Record Dates: First submitted 2006-02-21; First posted 2006-05-03 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Diphtheria; Hepatitis B; Poliomyelitis; Tetanus; Acellular Pertussis
MeSH Terms: conditions — Diphtheria; Hepatitis B; Poliomyelitis; Tetanus

INTERVENTIONS:
Biological: DTPa-HBV-IPV/Hib vaccine

SUMMARY:
In this study, infants will be randomly allocated into three groups:

* one group of subjects will receive DTPa-HBV-IPV/Hib vaccine (new formulation)
* the second group of subjects will receive DTPa-HBV-IPV/Hib vaccine (current formulation)
* the third group of subjects will receive DTPa-HBV-IPV vaccine The study will be double-blind for the two groups receiving the DTPa-HBV-IPV/Hib vaccine (new or current formulation). The study will be single-blind for the group receiving DTPa-HBV-IPV vaccine.

DETAILED DESCRIPTION:
A study to compare the immunogenicity & safety of 2 formulations of GlaxoSmithKline (GSK) Biologicals' DTPa-HBV-IPV/Hib vaccine given in healthy infants at 3,4 & 5 months age. The immunogenicity & safety of DTPa-HBV-IPV vaccine will also be evaluated in a 3rd group of subjects Subjects in the group that will receive DTPa-HBV-IPV/Hib vaccine (current formulation) will be the control group for the group that will receive DTPa-HBV-IPV/Hib vaccine (new formulation)

ELIGIBILITY:
"Inclusion criteria:

* A healthy male or female infant between, and including, 11 and 17 weeks of age at the time of the first vaccination.
* Infant born to known hepatitis B surface antigen (HBsAg) seronegative mother (documented laboratory result of HBsAg assay from the maternal blood sample is available).
* Born after a normal gestation period (between 36 and 42 weeks).
* Written informed consent obtained from the parent or guardian of the subject.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Any chronic drug therapy to be continued during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of study vaccine and ending 30 days after the last vaccine dose.
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B and/or Haemophilus influenzae diseases.
* Known history of or exposure to diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B and/or Haemophilus influenzae diseases since birth.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.

"

Ages: 11 Weeks to 17 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 415
Dates: Start 2006-04; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
One month after vaccination, measurement of antibodies against all vaccine antigens.

SECONDARY OUTCOMES:
Immunogenicity: One month after vaccination, vaccine response for the pertussis antigens.
Reactogenicity & safety: After each dose, solicited (day 0-3, local & general) & unsolicited (day 0-30) symptoms. Over the full course of the study: serious adverse events (SAEs)."

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Russia (3):
  - GSK Investigational Site, Murmansk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Syktyvkar

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 105910 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 105910 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105910 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105910 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105910 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105910 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register